CLINICAL TRIAL: NCT00831233
Title: A Randomised, Parallel-arm, Open-label Trial Comparing Degarelix With Goserelin Plus Anti-androgen Flare Protection (Bicalutamide), in Terms of Reduction in International Prostate Symptom Score (IPSS), in Patients With Lower Urinary Tract Symptoms (LUTS) Secondary to Locally Advanced Prostate Cancer
Brief Title: Symptomatic Study Investigating Degarelix in Patients Suffering From Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment due to rare targeted population
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS28; 2008-004338-26 (EudraCT Number)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Goserelin; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Degarelix 240 mg/80 mg (Experimental): Degarelix 240 mg (40 mg/mL) + 80 mg (20 mg/mL)
  Interventions: Drug: Degarelix
- Goserelin (3.6 mg) + bicalutamide (50 mg) (Active Comparator): Goserelin (3.6 mg) + bicalutamide (50 mg)
  Interventions: Drug: Goserelin; Drug: Bicalutamide

INTERVENTIONS:
Drug: Degarelix — The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The second and third doses of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections on Days 28 and 56, respectively.
  Other Names: FE200486
  Arms: Degarelix 240 mg/80 mg
Drug: Goserelin — Goserelin implants (3.6 mg) were inserted s.c. into the abdominal wall every 28 days. The second and third doses of goserelin were administered on Days 31 and 59, respectively.
  Other Names: Zoladex
  Arms: Goserelin (3.6 mg) + bicalutamide (50 mg)
Drug: Bicalutamide — On Day 0, three days before the first dose of goserelin on Day 3, patients began once-daily per-oral (p.o.) treatment with bicalutamide (50 mg) as anti-androgen flare protection; this treatment continued for 14 days after the first dose of goserelin.
  Other Names: Casodex
  Arms: Goserelin (3.6 mg) + bicalutamide (50 mg)

SUMMARY:
The purpose of this trial was to see how well a new trial drug (degarelix) worked on lower urinary tract symptoms (also known as LUTS) in prostate cancer patients as compared to how a standard drug hormonal treatment worked on the same symptoms. The advancement/worsening of prostate cancer may be associated with LUTS and the symptoms may impact the ability to urinate normally and thereby the quality of life for these patients.

Patients were randomly selected (like flipping a coin) to receive either degarelix or standard hormone therapy (combination of goserelin and bicalutamide) for a 3 month treatment period. During this period the relief of urinary symptoms was evaluated via a questionnaire filled in by patients and addressing the severity and frequency of their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent before any trial-related activity is performed
* Has a confirmed prostate cancer in which this type of treatment is needed.

Exclusion Criteria:

* Previous treatment for prostate cancer
* Previous trans-urethral resection of the prostate
* Current use of 5-alpha reductase inhibitor or α-adrenoceptor antagonist.
* Patients in need of external beam radiotherapy to be started at the same time as hormone therapy
* Certain risk factors for abnormal heart rhythms/QT prolongation (corrected QT interval over 450 msec., Torsades de Pointes or use of certain medications with potential risk)
* History of severe untreated asthma, anaphylactic reactions, or severe urticaria and/or angioedema.
* Hypersensitivity towards any component of the investigational product
* Other previous cancers within the last five years with the exception of prostate cancer and some types of skin cancer.
* Clinical disorders other than prostate cancer including but not limited to renal, haematological, gastrointestinal, endocrine, cardiac, neurological, psychiatric disease, alcohol or drug abuse or other conditionals as judged by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (33):
- Germany (10):
  - Facharztpraxis für Urologie, Bamberg
  - Gemeinschaftspraxis, Borken
  - Gemeinschaftspraxis, Cologne
  - Universitätsklinikum Dresden, Dresden
  - Euromed Clinic, Fürth
  - Urologische Gemeinschaftspraxis, Hamburg
  - VITURO Gesellschaft für Klinische Studien, Leipzig
  - Klinikum Offenbach GmbH, Offenbach
  - Urologische Klinik Planegg, Planegg
  - Wuppertaler Gemeinschaftspraxis, Wuppertal
- Spain (13):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Principe de Asturias, Alcalá de Henares-Madrid
  - Fundacion Hospital Alcorcón, Alcorcón
  - Fundación Puigvert, Barcelona
  - Hospital de Basurto, Bilbao (Bizkaia)
  - Hospital universitario Ramón y Cajal, Madrid
  - Hospital Clinico Universitario S. Carlos, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Manacor, Manacor
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Santiago de Compostela, Santiago de Compostela
  - Hospital Virgen Macarena, Seville
  - Hospital Xeral de Vigo, Vigo
- United Kingdom (10):
  - United Bristol Healthcare NHSTrust Bristol Royal Infirmary, Bristol
  - Falkirk and District Royal Infirmary, Falkirk
  - Southern General Hospital, Glasgow
  - Castle Hill Hospital, Hull
  - Whipps Cross University Hospital, London
  - The Royal Free Hospital, London
  - King's College Hospital, London
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield South, Sheffield
  - Sunderland Royal Hospital, Sunderland

REFERENCES:
- [Result] Anderson J, Al-Ali G, Wirth M, Gual JB, Gomez Veiga F, Colli E, van der Meulen E, Persson BE. Degarelix versus goserelin (+ antiandrogen flare protection) in the relief of lower urinary tract symptoms secondary to prostate cancer: results from a phase IIIb study (NCT00831233). Urol Int. 2013;90(3):321-8. doi: 10.1159/000345423. Epub 2012 Dec 15. PMID 23258223
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited by outpatient urologists. 280 participants were to be randomised in a 3:1 ratio to one of two treatment groups (210 patients were to be treated with degarelix; 70 patients were to be treated with goserelin plus bicalutamide). The trial was stopped early due to poor recruitment.
Period: Overall Study
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Started | 29 (Intention-to-treat (ITT) population.) | 13 (ITT population.)
Full Analysis Set (FAS) | 27 (2 participants were randomised but never treated.) | 13
Per Protocol (PP) Analysis Set | 26 | 11
Completed | 26 | 12
Not Completed | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Selection Criteria Not Met | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg) | Total
Number analyzed (Participants) | 27 | 13 | 40
Age Continuous [Mean (Standard Deviation); unit: years] — Full Analysis Set (FAS).
  years | 69.9 (8.68) | 71.0 (8.39) | 70.3 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants] — FAS.
  Participants
    Female | 0 | 0 | 0
    Male | 27 | 13 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants] — FAS.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 27 | 12 | 39
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — FAS.
  participants
    Spain | 4 | 4 | 8
    Germany | 13 | 7 | 20
    United Kingdom | 10 | 2 | 12
Body weight [Mean (Standard Deviation); unit: kilogram] — FAS.
  kilogram | 81.4 (14.0) | 78.2 (8.5) | 80.3 (12.5)
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter] — FAS.
  kilogram per square meter | 26.7 (4.06) | 26.8 (3.75) | 26.7 (3.91)
Gleason Score [Number; unit: participants] — FAS. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    2-4 | 0 | 0 | 0
    5-6 | 2 | 0 | 2
    7-10 | 25 | 13 | 38
Stage of Prostate Cancer [Number; unit: participants] — FAS. Prostate cancer stage was classified according to the Tumor, Nodes, and Metastatic (TNM) scale to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor. The majority of participants did not have their prostate cancer classified for the complete TNM scale (17 participants) or were known for having metastatic prostate cancer (14 participants).
  participants
    Localized | 4 | 0 | 4
    Locally Advanced | 4 | 1 | 5
    Metastatic | 10 | 4 | 14
    Not Classifiable | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total International Prostate Symptom Score (IPSS) at Week 12
Description: The IPSS is a tool commonly used to assess the severity of lower urinary tract symptoms (LUTS), and to monitor the progress of the disease once treatment has been initiated. The participant completes a questionnaire containing 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Each question is assigned a score of 0-5. The total score is then classified according to the following scale: 0 to 7 = mildly symptomatic; 8 to 19 = moderately symptomatic; and 20 to 35 = severely symptomatic.
Time Frame: After treatment of 12 weeks compared to Baseline
Population: Full Analysis Set (FAS) + Per Protocol (PP) Analysis Set, Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 27 | 13
score on scale | -11.2 (8.29) | -7.69 (7.61)
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); Estimates from analysis of variance with treatment and country as factors and age and baseline value as covariates; Test type: Non-Inferiority or Equivalence — The trial was positive if the treatment contrast of degarelix versus goserelin plus bicalutamide in adjusted (for baseline total IPSS, age, and country) mean change from baseline in total IPSS was statistically significantly smaller (two-sided at α=0.05 level) than Δ=3 points in both the FAS and the PP analysis set. If the Week 12 treatment assessment of IPSS was missing the LOCF approach was used, i.e., the IPSS closest to and before Week 12 was used; p = 0.1973, ANCOVA — FAS; The baseline score, age, and country were used as covariates and treatment was used as a factor in the analysis; Mean Difference (Final Values) = -2.95, 95% CI 2-sided [-7.51 to 1.61]
Statistical Analysis 2: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); Estimates from analysis of variance with treatment and country as factors and age and baseline value as covariates; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0398, ANCOVA — PP analysis set; The baseline score, age, and country were used as covariates and treatment was used as a factor in the analysis; Mean Difference (Final Values) = -5.88, 95% CI 2-sided [-11.5 to -0.291]

2. Secondary Outcome: Change From Baseline in Total IPSS at Weeks 4 and 8
Description: as for outcome 1
Time Frame: After treatment of 4 and 8 weeks compared to Baseline
Population: FAS, LOCF.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 26 | 13
score on scale
  Week 4 | -7.31 (5.83) | -4.62 (5.49)
  Week 8 | -9.46 (6.94) | -8.08 (9.00)
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); Week 4. Estimates from analysis of variance with treatment and country as factors and age and baseline value as covariates; Test type: Superiority or Other; p = 0.2298, ANCOVA; The baseline score, age, and country were used as covariates and treatment was used as a factor in the analysis for the FAS; Mean Difference (Final Values) = -2.47, 95% CI 2-sided [-6.58 to 1.64]
Statistical Analysis 2: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); Week 8. Estimates from analysis of variance with treatment and country as factors and age and baseline value as covariates; Test type: Superiority or Other; p = 0.6917, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.983, 95% CI 2-sided [-5.98 to 4.02]

3. Secondary Outcome: Change From Baseline in Maximum Urine Flow (Qmax) at Each Visit
Description: Uroflowmetry was used to quantify the maximum urine flow (Qmax; mL/sec)
Time Frame: After treatment of 4, 8 and 12 weeks compared to Baseline
Population: FAS, LOCF.
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 27 | 13
mL/sec
  Week 4 | 3.63 (7.82) | 3.55 (3.80)
  Week 8 | 4.74 (6.60) | 3.52 (3.58)
  Week 12 | 3.62 (7.37) | 2.07 (4.57)
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8151, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.553, 95% CI 2-sided [-5.33 to 4.22]
Statistical Analysis 2: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.455, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [-2.46 to 5.38]
Statistical Analysis 3: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); Week 12. Estimates from analysis of variance with treatment and country as factors and age and baseline value as covariates; Test type: Superiority or Other; p = 0.3186, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.02, 95% CI 2-sided [-2.04 to 6.08]

4. Secondary Outcome: Change From Baseline in Residual Volume (Vresidual) at Each Visit
Description: Uroflowmetry was used to quantify the residual volume (Vresidual; mL)
Time Frame: After treatment of 4, 8 and 12 weeks compared to Baseline
Population: FAS, LOCF.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 27 | 13
mL
  Week 4 | -36.2 (148) | -19.8 (63.5)
  Week 8 | -43.8 (133) | -19.6 (85.4)
  Week 12 | -50.7 (135) | -13.4 (85.8)
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5627, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 15.2, 95% CI 2-sided [-37.8 to 68.2]
Statistical Analysis 2: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.8284, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 5.91, 95% CI 2-sided [-49.1 to 60.9]
Statistical Analysis 3: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.5984, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 12.2, 95% CI 2-sided [-34.4 to 58.8]

5. Secondary Outcome: Change From Baseline in Prostate Size Based on Trans Rectal Ultra Sound (TRUS) at Week 12
Description: TRUS is a method of measuring the size of the prostate.
Time Frame: After 12 weeks treatment compared to Baseline
Population: FAS, Observed Cases (OC).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 26 | 11
mL | -22.4 (14.8) | -13.4 (10.0)
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); Estimates from analysis of variance with treatment and country as factors and age and baseline value as covariates; Test type: Superiority or Other; p = 0.1018, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -7.83, 95% CI 2-sided [-17.3 to 1.64]

6. Secondary Outcome: Number of Participants With Testosterone <=0.5 Nanograms/Milliliter at Each Visit
Time Frame: After treatment of 4, 8 and 12 weeks compared to Baseline
Population: FAS, OC.
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 27 | 13
participants
  Week 4 | 26 | 12
  Week 8 | 25 | 12
  Week 12 | 27 | 12

7. Secondary Outcome: Percentage Change From Baseline in Prostate-specific Antigen (PSA) Concentration at Each Visit
Time Frame: After treatment of 4, 8 and 12 weeks compared to Baseline
Population: FAS, LOCF.
Measure: Median (Full Range); unit: percentage
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 27 | 12
percentage
  Week 4 | -85.72 [-97.87 to 234.97] | -93.44 [-98.33 to -87.09]
  Week 8 | -89.2 [-99.47 to -31.62] | -97.26 [-99.72 to -87.56]
  Week 12 | -93.87 [-99.83 to -64.71] | -97.78 [-99.72 to -94.52]

8. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Related to Urinary Symptoms at Each Visit
Description: The IPSS questionnaire included an additional single question to assess the participant's QoL in relation to his urinary symptoms. The question was: 'If you were to spend the rest of your life with your urinary condition the way it is now, how would you feel about that?' The possible answers to this question ranged from 'delighted' (a score of '0') to 'terrible' (a score of '6'). The figures in the tables present the change (ie decrease) in IPSS QoL score, i.e. the bigger the decrease the better QoL.
Time Frame: After treatment of 4, 8 and 12 weeks compared to Baseline
Population: FAS, OC.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 27 | 13
score on scale
  Week 4 | -0.96 (0.92) | -0.54 (1.51)
  Week 8 | -1.54 (1.42) | -0.73 (2.20)
  Week 12 | -1.77 (1.73) | -0.55 (1.69)

9. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight. The table presents the number of participants with normal baseline and at least one post-baseline markedly abnormal value.
Time Frame: Baseline to 12 weeks of treatment
Population: FAS. One participant in the degarelix group did not have any assessment of vital signs or body weight (the number of participants in this group is thus 26).
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 26 | 13
participants
  Diastolic blood pressure <=50 and decrease >=15 | 0 | 0
  Diastolic blood pressure >=105 and increase >=15 | 0 | 0
  Systolic blood pressure <=90 and decrease >=20 | 0 | 0
  Systolic blood pressure >=180 and increase >=20 | 0 | 0
  Heart rate <=50 and decrease >=15 | 0 | 0
  Heart rate >=120 and increase >=15 | 0 | 0
  Body weight decrease of >=7 percent | 1 | 0
  Body weight increase of >=7 percent | 1 | 0

10. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Safety Laboratory Variables
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) levels of safety laboratory variables. Only the laboratory variables that had at least on participant with one abnormal value are presented, many more variables were included in the trial.
Time Frame: Baseline to 12 weeks of treatment
Population: FAS.
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 27 | 13
participants
  B-Haematocrit (Ratio) <=0.37 | 5 | 1
  B-Platelet count (10^9/L) <=75 | 1 | 0
  S-Calcium (mmol/L) <=1.8 | 1 | 0
  S-Potassium (mmol/L) >=5.8 | 0 | 1
  S-Urea nitrogen (mmol/L) >=10.7 | 1 | 2

ADVERSE EVENTS:
Time Frame: 12 weeks.
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/13
Other Adverse Events (participants affected / at risk) | 14/27 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240 mg/80 mg (N=27) | Goserelin (3.6 mg) + Bicalutamide (50 mg) (N=13)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240 mg/80 mg (N=27) | Goserelin (3.6 mg) + Bicalutamide (50 mg) (N=13)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Reproductive tract hypoplasia, male (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Injection site pain (General disorders) | 6 (16) | 0 (0)
Injection site erythema (General disorders) | 3 (5) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 3 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 3 (3) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.